CLINICAL TRIAL: NCT03294902
Title: Improving Radiological Outcomes in Arterial Disease - A Pilot Evaluation of the Pedra Tissue Perfusion Monitoring System
Acronym: IROAD
Status: Completed | Type: Observational
Sponsor: Pedra Technology, PTE LTD (Industry)
Responsible Party: Sponsor
Other Study IDs: CIP-01
Record Dates: First submitted 2017-08-25; First posted 2017-09-27 (Actual); Last update posted 2020-09-21 (Actual); Status verified 2020-09

CONDITIONS: Peripheral Arterial Disease; Chronic Limb Ischemia
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Critical Limb Ischaemia (CLI) Group with tibial arterial dis: Up to 20, but at least 8 subjects with a Rutherford grade 4 or 5 critically ischemic foot, where the primary intention is to treat at least one occluded tibial vessel or 2 severely stenosed tibial vessels. The treatment of SFA stenoses of less than 70%, as confirmed by duplex or CT, is acceptable in parallel in this group.
  Interventions: Device: Pedra Tissue Perfusion Monitor
- Peripheral Artery Disease (PAD) Group with SFA disease: Up to 20, but at least 8 subjects with a clinical diagnosis of claudication and duplex or CT-confirmed SFA stenoses greater than 70%, with no intention of primarily treating any tibial disease at this encounter.
  Interventions: Device: Pedra Tissue Perfusion Monitor
- PAD-free group (Healthy Volunteer Group): Up to 20 subjects with no clinical diagnosis of peripheral vascular disease.
  Interventions: Device: Pedra Tissue Perfusion Monitor

INTERVENTIONS:
Device: Pedra Tissue Perfusion Monitor — This study is a prospective single-centre, device observational study designed to enroll up to 60 evaluable subjects at 1 investigational site in the United Kingdom. Eligible subjects, who meet the requirements for one of the 3 distinct subject groups: (1) Critical Limb Ischaemia group, (2) Peripheral artery disease with superficial femoral arterial (SFA) or popliteal artery disease and (3) PAD-free group. Subjects who meet study eligibility criteria will be enrolled consecutively until the total number of subjects is enrolled per each group as outlined in the protocol. All subjects at the investigational site will be enrolled in the presence of a member of the Sponsor or selected designee in order to assist with the device operation and to verify that all protocol assessments are completed appropriately at baseline.

SUMMARY:
The Pedra Technologies' PedraTM device is a non-invasive, diagnostic device intended to measure foot perfusion by assessing blood flow. The PedraTM device comprises a compact instrument console connected to a sensor that is pasted onto the patient's foot during perfusion assessment. Through skin contact, the device is able to monitor tissue perfusion at depths of up to 7.5mm. The monitor console contains opto-electronic instrumentation including coherent infrared light sources, photo detectors, and display/control electronics. The sensor comprises passive fiber-optic conduits, which transfer infrared light from the console to the patient, and relays scattered light from the patient back to the console. The intensity of light emitted from the sensor is less than 3 mW, well within the safety envelope of Class I laser systems and comparable (or lower than) other commercially available devices such as laser Doppler systems. The sole point of contact with the patient is a layer of medical grade adhesive tape, which is used to paste the flat sensor onto intact skin.

ELIGIBILITY:
General Inclusion Criteria:

1. The patient is a male or non-pregnant female ≥ 40 to 90 years of age
2. The patient is willing to comply with protocol-specified follow-up evaluations
3. The patient has been informed of the nature of the study, agrees to its provisions and has willingly provided written informed consent, approved by the appropriate Ethics Committee (EC)

Cohort Specific Inclusion Criteria:

Critical Limb Ischaemia Group Inclusion Criteria:

1. The subject is referred for a percutaneous peripheral revascularisation procedure on one of their lower limbs within 2 weeks of Baseline assessments.
2. Rutherford grade 4 or 5 critically ischemic foot, where the primary intention is to treat at least one occluded tibial vessel or 2 severely stenosed tibial vessels.

Peripheral Arterial Disease Group Inclusion Criteria:

1. The subject is referred for a percutaneous peripheral revascularisation procedure on one of their lower limbs within 2 weeks of Baseline assessments.
2. This subject must have a clinical diagnosis of claudication and duplex or CT-confirmed SFA or popliteal artery stenoses greater than 70%, with no intention of primarily treating any tibial disease at this encounter.

PAD-Free Group Inclusion Criteria:

1. The subject is recruited voluntarily
2. Absence of peripheral vascular disease determined by questionnaire and clinical review (triphasic signals on hand-held Doppler)

Exclusion Criteria:

1. Infusion of vasoactive medications within the past 24 hours
2. The presence of a known chronic history of anaemia (i.e. Hb <8g/dL)
3. Congestive heart failure defined by NYHA Classification 3 or 4
4. The absence of intact skin at suitable measurement sites on the foot.
5. The presence of invasive soft tissue infection in the toes spreading into the forefoot.
6. The presence of physical impediment to the method of measurements being completed (i.e. absent first two toes, extensive ulceration, excessive oedema, pressure dressings or heavy bandaging, etc.)
7. The presence of a non-salvageable foot or a Rutherford 6 wound.
8. The presence of other conditions, which in the opinion of the Investigator, may compromise the subject safety or comfort.
9. The presence of other conditions, which in the opinion of the Investigator, may compromise the accuracy of the data obtained.
10. The patient is a vulnerable or protected adult, or is unable to provide consent.
11. The patient is unable to comply with the measurement protocol.
12. Pregnant subjects

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The 3 distinct subjects groups are divided as such:
  * Critical Limb Ischaemia (CLI) Group with tibial arterial disease: Up to 20, but at least 8 subjects with a Rutherford grade 4 or 5 critically ischemic foot, where the primary intention is to treat at least one occluded tibial vessel or 2 severely stenosed tibial vessels. The treatment of SFA stenoses of less than 70%, as confirmed by duplex or CT, is acceptable in parallel in this group.
  * Peripheral Artery Disease (PAD) Group with SFA disease: Up to 20, but at least 8 subjects with a clinical diagnosis of claudication and duplex or CT-confirmed SFA stenoses greater than 70%, with no intention of primarily treating any tibial disease at this encounter.
  * PAD-free Group (Healthy Volunteer Group): Up to 20 subjects with no clinical diagnosis of peripheral vascular disease.
Sampling Method: Non-Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2018-05-30 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Baseline safety endpoint: The absence of immediately observable skin reaction (rash; local oedema, blistering of the skin) in ≥ 90% of subjects after removal of the Pedra sensors. | Baseline visit: 30-60 minutes after pad removal
  This observation assessment is completed by the physician post removal of the adhesive pads. It is either a "yes" or a "no" in observing if there is a skin reaction to the adhesive pads when they are removed from the skin and also documentation of what type of reaction (rash; local oedema, blistering of the skin).
During procedure safety endpoint: The absence of immediately observable skin reaction (rash; local oedema, blistering of the skin) in ≥ 90% of subjects after removal of the Pedra sensors. | During procedure visit: 30-60 minutes after pad removal
  This observation assessment is completed by the physician post removal of the adhesive pads. It is either a "yes" or a "no" in observing if there is a skin reaction to the adhesive pads when they are removed from the skin and also documentation of what type of reaction (rash; local oedema, blistering of the skin).
36-hrs post-procedure/ discharge visit safety endpoint: The absence of immediately observable skin reaction (rash; local oedema, blistering of the skin) in ≥ 90% of subjects after removal of the Pedra sensors. | 36-hrs post-procedure/ discharge visit: 30-60 minutes after pad removal
  This observation assessment is completed by the physician post removal of the adhesive pads. It is either a "yes" or a "no" in observing if there is a skin reaction to the adhesive pads when they are removed from the skin and also documentation of what type of reaction (rash; local oedema, blistering of the skin).

CONTACTS AND LOCATIONS:
Locations (1):
- Addenbrooke's Hospital, Department of Vascular Surgery, Cambridge, United Kingdom

IPD SHARING:
Plan to Share IPD: No